CLINICAL TRIAL: NCT01740323
Title: Meriva for Treatment-induced Inflammation and Fatigue in Women With Breast Cancer
Brief Title: Phase II Study of Curcumin vs Placebo for Chemotherapy-Treated Breast Cancer Patients Undergoing Radiotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Andrew H Miller (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Andrew H Miller, Sponsor Investigator, Emory University
Organization: Emory University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00055328; Winship2139-11 (Other: Other); R21CA178603 (NIH)
Record Dates: First submitted 2012-11-30; First posted 2012-12-04 (Estimated); Results first posted 2019-09-18 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Chemotherapy; Radiotherapy; NF-kB; DNA Binding; Curcumin; IL-6; TNF; sTNFR2; IL-1-ra; Fatigue; Cytokine
MeSH Terms: conditions — Breast Neoplasms; Fatigue | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Curcumin (Experimental): 500 mg BID
  Interventions: Drug: Curcumin

INTERVENTIONS:
Drug: Placebo — daily placebo for 6 weeks
  Arms: Placebo
Drug: Curcumin — 500 mg BID
  Other Names: Meriva
  Arms: Curcumin

SUMMARY:
The main purpose of the investigation is to determine if curcumin reduces NF-kB DNA binding and ultimately its downstream mediator IL-6 in patients receiving XRT for their breast cancer after having completed chemotherapy. Patients who have received prior chemotherapy will be eligible, because we have found that this enriched population is at particular risk for exhibiting increased NF-kB DNA binding and IL-6 following XRT.

DETAILED DESCRIPTION:
As many as 60% of breast cancer (BrCA) patients receiving radiation are known to develop fatigue with about 30% suffering persistent fatigue several months to years after treatment completion (12-23). The physical, psychological, and molecular mechanisms by which patients develop fatigue are poorly understood and most likely multi-factorial. One pathway that has received considerable attention is nuclear factor-kappa B (NF-kB)(24). The NF-kB pathway has emerged as having an important role not only in cancer treatment resistance but in the development of fatigue. NF-kB activation leads to over expression of interleukin (IL)-1beta, IL-6, and tumor necrosis factor (TNF)-alpha, all factors related to inflammation and factors that have been found to be upregulated in patients receiving radiation as well as BrCA survivors with fatigue (25-29). A recently published study looking at TNF-alpha, fatigue and cachexia in cancer patients receiving docetaxol showed that NF-kB is upregulated in fatigued patients and that agents which inhibit TNF-alpha lead to better tolerance of chemotherapy dose escalation (30). Work by our group and others has shown that ionizing radiation increases NF-kB pathway activity in circulating immune cells (as well as within breast cancer cells) and that this effect is most pronounced in women previously treated with chemotherapy (31, 32). Our work has shown that the NF-kB pathway activity in circulating immune cells is also related to fatigue development in BrCA patients treated with radiation and that patients most at risk for persistent fatigue and NF-kB pathway activity are those who have received chemotherapy for their breast cancer (31).

Curcumin, a known inhibitor of NF-kB, has been shown to decrease NF-kB activation in human participants. In a recent study, 8 grams of curcumin by mouth daily for 8 weeks was well tolerated in patients with pancreatic cancer and other pre-malignant conditions with no associated toxicities (6, 8). Although there is concern over the body's absorption of curcumin, the bioavailability of curcumin in the study of pancreatic cancer patients was shown, with peak drug levels at 22 to 41ng/mL that remained relatively constant over the first 4 weeks of treatment with 8 grams of curcumin daily (8). Clinical trials with daily dosages of 1,125 to 2,500mg have also confirmed the safety of curcumin and also shown its ability to decrease inflammation in patients with rheumatoid arthritis and in post-operative patients (6, 33, 34). In vivo murine models of chronic fatigue syndrome have also shown that curcumin may also alleviate symptoms of fatigue (35). While these studies are promising, very little is known about the capacity of Meriva to inhibit NF-kB in women treated for BrCA. We hypothesize that oral Meriva, a known inhibitor of NF-kB, may be used to decrease levels of NF-kB activity in BrCA patients previously treated with chemotherapy who go on to receive radiotherapy (XRT), a carefully chosen group of patients at particular risk for high levels of NF-kB DNA binding (a direct measure of NF-kB pathway activity).

We have chosen to administer oral Meriva, 500mg BID, in our patient population based on the above data. Meriva-500 is a curcumin formulation that also contains phosphatidylcholine, derived from soy that has been shown to aid in absorption of curcumin (9), permitting a lower overall dose of curcumin. Of note, 1000 mg Meriva contains 200 mg curcuminoids (>90% curcumin).

By decreasing activity of NF-kB and ultimately plasma IL-6, fatigue may improve in BrCA patients taking Meriva. Results from this study will contribute to the limited research available on the capacity of curcumin treatment, including Meriva, to inhibit NF-kB activation in vivo as well as symptoms of fatigue associated with excessive NF-kB pathway activity in BRCA patients.

ELIGIBILITY:
Inclusion Criteria:

* Female breast cancer patients over the age of 18 will be recruited for this study. Patients enrolled in the study will meet standard criteria for whole breast XRT.

Exclusion Criteria:

* Subjects will be excluded for a number of medical conditions that are contraindications to XRT and/or might confound the relationship among fatigue, and inflammation, including pregnancy, major psychiatric disorders, autoimmune or inflammatory disorders, chronic infectious diseases (e.g. HIV, hepatitis B or C), neurologic disorders and uncontrolled cardiovascular, metabolic, pulmonary or renal disease (as determined by medical history, physical examination and laboratory testing). Subjects with a history of a major psychiatric disorder including Schizophrenia or Bipolar Disorder or a diagnosis of Substance Abuse or Dependence within the past 1 year (as determined by standardized psychiatric interview) will be excluded. Subjects taking drugs known to affect the immune system (e.g. glucocorticoids, methotrexate) will also be excluded. Subjects using supplements or other natural products with one week of starting medications, excluding vitamins and calcium supplementation or at the discretion of the attending physician, will be excluded. Patients who have evidence of infection as determined by history, physical exam or laboratory testing (complete blood count and urinalysis) at baseline will be excluded. In addition, patients who develop evidence of infection (as determined by history, physical exam or laboratory testing) during the study will be discontinued from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-05; Primary Completion 2018-07-27 (Actual); Study Completion 2018-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew H Miller, MD, Principal Investigator — Emory Winship Cancer Institute
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Curcumin
Started | 15 | 15
Completed | 13 | 15
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Randomized but did not take study drug | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Curcumin | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.87 (10.67) | 50.47 (10.01) | 51.17 (10.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 15 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 6 | 13
  White | 7 | 7 | 14
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: PBMC NF-kB DNA Binding Measured in ng/Well
Description: The primary outcome to be measured will be the change in NF-kB DNA binding (measured in peripheral blood mononuclear cells as ng/well) after six weeks of treatment with daily placebo or Meriva. NF-kB DNA binding and has been associated with fatigue in breast cancer patients.
Time Frame: Baseline, 6 weeks following completion of XRT
Measure: Mean (Standard Deviation); unit: ng/well
Arm/Group | Placebo | Curcumin
Number analyzed (Participants) | 13 | 15
ng/well
  Baseline | 9.01 (14.70) | 9.56 (5.63)
  6 weeks post-treatment | 17.54 (9.24) | 16.04 (16.13)

2. Primary Outcome: Plasma TNF-alpha
Description: The secondary outcome to be measured will be the change in plasma TNF-alpha after six weeks of treatment with daily placebo or Meriva. Plasma TNF-alpha is a downstream mediator of NF-kB DNA binding and has been associated with fatigue in breast cancer patients.
Time Frame: Baseline, 6 weeks following completion of XRT
Measure: Mean (Standard Deviation); unit: ng/well
Arm/Group | Placebo | Curcumin
Number analyzed (Participants) | 13 | 15
ng/well
  Baseline | 5.87 (3.52) | 4.93 (1.75)
  6 weeks post-treatment | 4.93 (1.75) | 5.24 (0.97)

3. Primary Outcome: Plasma sTNFR2 Measured in pg/ml
Description: The secondary outcome to be measured will be the change in plasma sTNFR2 (in pg/ml) after six weeks of treatment with daily placebo or Meriva. Plasma sTNFR2 is a downstream mediator of NF-kB DNA binding and has been associated with fatigue in breast cancer patients.
Time Frame: Baseline, 6 weeks following completion of XRT
Population: Assays were not analyzed due to lack of funding.
Arm/Group | Placebo | Curcumin
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Plasma IL-1ra Measured in pg/ml
Description: The secondary outcome to be measured will be the change in plasma IL-1ra (in pg/ml) after six weeks of treatment with daily placebo or Meriva. Plasma IL-1ra is a downstream mediator of NF-kB DNA binding and has been associated with fatigue in breast cancer patients.
Time Frame: Baseline, 6 weeks following completion of XRT
Population: Assays were not analyzed due to lack of funding.
Arm/Group | Placebo | Curcumin
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Plasma IL-6 Measured in pg/ml
Description: The primary outcome to be measured will be the change in plasma IL-6 after six weeks of treatment with daily placebo or Meriva.
Time Frame: Baseline, 6 weeks following completion of XRT
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | Curcumin
Number analyzed (Participants) | 13 | 15
pg/mL
  Baseline | 2.29 (3.26) | 1.84 (1.32)
  6 weeks post-treatment | 2.04 (2.36) | 1.77 (1.59)

6. Primary Outcome: Plasma C-reactive Protein (CRP) Measured in mg/L
Description: The primary outcome to be measured will be the change in plasma CRP after six weeks of treatment with daily placebo or Meriva.
Time Frame: Baseline, 6 weeks following completion of XRT
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Placebo | Curcumin
Number analyzed (Participants) | 13 | 15
mg/L
  Baseline | 2.71 (2.97) | 2.72 (3.48)
  6 weeks post-treatment | 3.85 (4.36) | 2.30 (2.95)

7. Secondary Outcome: Fatigue
Description: The secondary outcome to be measured will be the change in fatigue (as measured by the Multidimensional Fatigue Inventory [MFI] total score) after six weeks of treatment with daily placebo or Meriva. The MFI is a 20-item scale designed to evaluate fatigue. Respondents use a scale ranging from 1 to 5 for each item to indicate how statements regarding fatigue represent their experiences. The range of scores is from a minimum of 20 and a maximum of 100. Higher total scores correspond with more acute levels of fatigue.
Time Frame: Baseline, 6 weeks following completion of XRT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Curcumin
Number analyzed (Participants) | 13 | 15
score on a scale
  Baseline | 56.69 (15.70) | 57.40 (13.30)
  6 weeks post-treatment | 50.23 (13.86) | 46.67 (13.62)

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: Events were assessed during weekly telephone calls with participants while they were on the study protocol. All adverse events were collected using the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0.
Arm/Group | Placebo | Curcumin
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 2/15
Other Adverse Events (participants affected / at risk) | 12/15 | 13/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=15) | Curcumin (N=15)
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1)
Motor vehicle accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=15) | Curcumin (N=15)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal symptoms (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 5 (5)
Sore/itchy throat (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Muscle pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 0 (0)
Fractured elbow (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (6)
Cold sore (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Blisters (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail loss (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Reflux/Indigestion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomach Pain (Gastrointestinal disorders) | 3 (3) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (4) | 5 (7)
Stool change/Flatulence (Gastrointestinal disorders) | 5 (5) | 3 (3)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1)
Menstrual changes (Reproductive system and breast disorders) | 4 (4) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast discomfort/pain (Reproductive system and breast disorders) | 3 (3) | 1 (1)
Headache (General disorders) | 5 (5) | 3 (5)
Vertigo/ Dizziness (General disorders) | 0 (0) | 2 (3)
Toothache (General disorders) | 1 (1) | 0 (0)
Chills/Hot flashes (General disorders) | 4 (4) | 4 (4)
Heart murmur/Palpitations (Cardiac disorders) | 0 (0) | 2 (2)
High Blood pressure (Cardiac disorders) | 0 (0) | 1 (4)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 1 (1)
Insomnia (Nervous system disorders) | 1 (1) | 3 (3)
Anxiety/Irritability/Mood change (Nervous system disorders) | 1 (1) | 3 (3)
Neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Carpal tunnel (Nervous system disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 2 (2)
Swollen Glands (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-22): https://cdn.clinicaltrials.gov/large-docs/23/NCT01740323/Prot_SAP_000.pdf